CLINICAL TRIAL: NCT05332535
Title: Effect Of Serious Game-Based Web Application On Stoma Care Education For Nursing Students
Brief Title: Serious Game On Stoma Care Education For Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Nursen Kulakac, Lecturer, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GumushaneU
Record Dates: First submitted 2021-12-14; First posted 2022-04-18 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Surgical Stoma; Nursing; Video Games
Keywords: Education; Nursing; Student; Surgical stoma; Video games

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious game web aplication (Experimental): Nursing students played the serious game for two weeks.
  Interventions: Behavioral: serious game based web application education
- Control grup (No Intervention)

INTERVENTIONS:
Behavioral: serious game based web application education — serious game based web application education for nursing students
  Arms: Serious game web aplication

SUMMARY:
Today, rapidly developing technology needs to be integrated into teaching environments and reconstructed teaching environments. When virtual reality applications, which are among the popular and innovative technologies, are examined, it is seen that participants are used in many areas of education. In this randomized controlled study, it was aimed to evaluate the impact of stoma care education by designing a serious game based web application that enables nursing students to gain skills and practice in psychomotor applications. The universe of the study will be students enrolled in the Surgical Diseases Nursing course in the spring semester of the 2020-2021 academic year at the Faculty of Health Sciences, Gümüşhane University. Students will be divided into two groups as control and experiment by randomization method. The data will be collected through introductory features form, 'Stoma Care Information Form', 'Stoma Care Skill Checklist' and Computer System Usability Survey. In the first stage of the study, the students will be given a 'Stoma Care Information Form' (first knowledge). 'Stoma Care Information Form' (second information) and 'Stoma Care Skill Checklist' will be applied after completing the theoretical lesson of stoma care and group work in the laboratory of students in the experimental and control groups. Unlike the control group, of students in the experimental group; A serious game-based web application on stoma care prepared as a support for formal education will be installed. After four weeks of the students attending formal education, 'Stoma Care Information Form' (third knowledge) and 'Stoma Care Skill Checklist' (second skill) will be applied. In the experiment and control group, two weeks later, the "Stoma Care Information Form" (fourth information) and "Stoma Care Skill Checklist" (third skill) will be applied again to test the permanence of the methods. Skill measurements of students will be made with an objective structured clinical exam. The results obtained after the application will be analyzed and the impact of serious game based web application on stoma care education will be determined

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in the HEMSEC-217 Emergency Nursing course for the first time,
* Having successfully completed the Internal Medicine Nursing course,
* He voluntarily agreed to participate in the study.
* Having internet access

Exclusion Criteria:

* To have received training (in-service training, course, seminar, etc.) on stoma care,
* Having graduated from a health vocational high school and having experience in stoma care,
* Taking the HEMSEC-217 Emergency Nursing course for the second time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
To measure nursing student's information | 4 week
  The data will be collected through introductory features form, 'Stoma Care Information Form', In the first stage of the study, the students will be given a 'Stoma Care Information Form' (first knowledge). 'Stoma Care Information Form' (second information) will be applied after completing the theoretical lesson of stoma care and group work in the laboratory of students in the experimental and control groups. There are 20 questions on the subject in the knowledge test and the lowest 0 and the highest 20 points are taken from the test. Increasing score indicates higher achievement.

SECONDARY OUTCOMES:
To measure nursing student's skill | 4 week
  Unlike the control group, the mobile phones of students in the experimental group; A serious game-based virtual reality mobile application on stoma care prepared as a support for formal education will be installed. After the students play the application, skill measurements will be made in the laboratory with 'Skill Checklists'. Skill measurements of students will be made with an objective structured clinical exam.The skill checklist includes 36 process steps that students are expected to perform. 2 points were given for each correct step evaluated in the list, 1 point for the missing step, and 0 points for each unfulfilled step. A minimum of 0 and a maximum of 72 points can be obtained from the skill checklist. Increasing score indicates higher achievement.

OTHER OUTCOMES:
To determine permanence of the method | 4 week
  The results obtained after the application will be analyzed and the impact of serious game based virtual reality mobile application on stoma care education will be determined. The scale consists of three sub-dimensions as system usefulness (items 1-6), quality of information (items 7-9), and interface quality (items 10-12), and item 13 measures overall satisfaction. Each item is scored as 1 (Strongly agree) - 7 (Strongly disagree). A low score from the scale indicates high usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Nurşen Kulakaç, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available 01.06.2022 and 01.12.2020
Access Criteria: Non